CLINICAL TRIAL: NCT02524015
Title: Novel Treatment For Pusher Syndrome Using Physical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Mary Kim, Assistant Professor, Residency Program Director, PM&R, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5150231
Record Dates: First submitted 2015-08-07; First posted 2015-08-14 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Pusher Syndrome
Keywords: stroke; pusher syndrome; contraversive pushing; lateropulsion; rehabilitation; physical therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Standard Physical Therapy
  Interventions: Other: Standard physical therapy
- Intervention (Experimental): Novel Physical Therapy
  Interventions: Other: Novel physical therapy

INTERVENTIONS:
Other: Novel physical therapy
  Arms: Intervention
Other: Standard physical therapy
  Arms: Control

SUMMARY:
The purpose of this study is to see if a specific physical therapy intervention speeds recovery from stroke-related "pusher syndrome."

ELIGIBILITY:
Inclusion Criteria:

* Recent (within 2 months) unilateral stroke
* Burke Lateropulsion Scale ≥ 2
* Age 21 to 89 years
* Ability to provide informed consent
* English-speaking

Exclusion Criteria:

* Prior stroke within the past 6 months
* Cerebellar stroke
* Stroke-related brain imaging (MRI or CT) unavailable
* Global or receptive aphasia
* Prior documented neurologic disorder (e.g., multiple sclerosis, Parkinson's)

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Recovery from pusher syndrome as measured by changes in the Burke Lateropulsion Scale score over time. | Initial, and then weekly until discharge from inpatient rehabilitation unit. Average inpatient stay is expected to be no greater than 4 weeks.
  The Burke Lateropulsion Scale (BLS) is used in the literature to measure the presence of pusher syndrome. We will measure BLS upon admission and at weekly intervals to monitor whether patients in the experimental group demonstrate faster recovery than the control group, as demonstrated by change in BLS score over change in time (days).